CLINICAL TRIAL: NCT06641739
Title: Comparative Clinical Trials of Laser Photobiomodulation and Platelets Rich in Growth Factors (PRGFs)-Assisted Flap Surgery in Treating Stage III Periodontal Defects: an In-Depth Analysis of Clinical Outcomes and Healing Processes
Brief Title: Photobiomodulation and Platelets Rich in Growth Factors (PRGFs)-Assisted Flap Surgery in Treating Stage III Periodontal Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nashwa Helaly Mohamed, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: laser and PRF in periodontitis
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Periodontal Diseases
Keywords: photobiomodulation; laser therapy; PRF; stage III periodontal diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Group 1: Ten patients will be treated with simplified papilla preservation flap with platelet-rich fibrin grafted into the defect site.
  Group 2: Ten patients will be treated the simplified papilla preservation flap with laser therapy performed into the defect site. The laser used in the study is diode lasers (940nm), with an output power of 3 W in the contact mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- • Laser-treated group (Active Comparator): Ten patients will be treated the simplified papilla preservation flap with laser therapy performed into the defect site. The laser used in the study is diode lasers ( 940nm), with an output power of 3 W in the contact mode.
  Interventions: Device: laser assisted SPPF
- platelets Rich Fibrin Graft (Active Comparator): Ten patients will be treated with simplified papilla preservation flap with platelet-rich fibrin grafted into the defect site.
  Interventions: Procedure: Platelet Rich Plasma

INTERVENTIONS:
Device: laser assisted SPPF — A full-thickness flaps were elevated. In the test sites after the SPPF access will be performed, root surface debridement will be meticulously performed, followed by intra-marrow penetrations (IMPs), on the defect walls using a 0.25 mm wide half round bur, mounted on a slow-speed handpiece. Following this, low-level laser biostimulation of the defect will be effected with an 940 nm diode laser at 3 W power, with an uninitiated 0.6mm optical fiber tip. The defects will be irradiated for 20 seconds in a continuous noncontact mode and then retracted for 8 seconds. This will be repeated for 3 times so that the defects were effectively lased for about 60 seconds.
  Arms: • Laser-treated group
Procedure: Platelet Rich Plasma — In the second group, following the SPPF, the defect will grafted with particulated PRF, which will be overlaid with a PRF membrane, without any adjunctive defect management measures. PRF will be prepared by collecting Intra-venous blood (from the antecubital vein) in a 10-ml sterile glass tube without anticoagulant and immediately centrifuged in a centrifugation machine at 3000 rpm for 10 minutes. It will result in the separation of blood into a structured fibrin matrix in the middle of the tube, just between the red corpuscles at the bottom and acellular plasma (platelet poor plasma) at the top. PPP will be discarded. PRF will be easily separated from the red corpuscles base using sterile tweezers and scissors.
  Arms: platelets Rich Fibrin Graft

SUMMARY:
Stage 3 periodontitis is a condition marked by swift and severe destruction of periodontal tissues. To effectively regenerate osseous defects resulting from periodontal disease, it is crucial to leverage the intrinsic regenerative potential of the periodontium via meticulously formulated therapeutic strategies

DETAILED DESCRIPTION:
The main treatment methods of periodontal diseases involve scaling and root planning (SRP), and periodontal surgery. Periodontopathogens, can penetrate deep by crossing the epithelial barrier which may be difficult to be remove by nonsurgical periodontal therapy (NSPT) alone. A multitude of grafted and non-grafted approaches have been used in the management of Intra-bony defects. However, they do not provide predictable periodontal regeneration.

A systematic review on the use of platelet-rich fibrin (PRF) for managing periodontal defects highlights its promising potential in periodontal regeneration. It forms a fibrin matrix that promotes angiogenesis and enhances healing at defected sites. The review emphasizes PRF's ability to sustain the release of growth factors, which are crucial for osteoblastic proliferation, migration, and adherence. This makes PRF an effective scaffold for cellular elements, facilitating periodontal tissue regeneration.

Laser photobiomodulation (PBM) has emerged as a promising adjunctive treatment as it stimulates cellular processes, enhancing the natural regenerative capabilities of periodontal tissues. Recent studies have demonstrated that PBM, particularly with diode, significantly improves clinical outcomes when combined with conventional periodontal treatments. It promotes osteoblastic proliferation, migration, and adherence, thereby facilitating bone regeneration and reducing periodontal pocket depth. Additionally, PBM enhances angiogenesis and modulates the release of growth factors, creating an optimal healing environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PPD =5 mm and clinical attachment loss of ≥3 mm;
* Presence of 2 walled or 3 walled infra-bony defects posterior segments;
* Evidence of ≥3 mm of intra-bony defect depth evaluated by the visualization of peri-apical radiographs.

Exclusion Criteria:

* Patients requiring antibiotic prophylaxis before the periodontal examination;
* Patients diagnosed with malocclusion at the site of the defect;
* Patients with systemic disease and/or on drugs that contraindicate periodontal surgery;
* Patients with a history of smoking and pan chewing;
* Sites with advanced class II & III furcation involvement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
-Evaluation of the changes in the clinical attachment loss | [Time Frame: at base line, 1 month and 3 months after treatment]
  Attachment level will be measured using UNC15(University of North Carolina) periodontal probe. Clinical attachment loss will be measured as the distance from the cemento-enamel junction to the base of the pocket.[Time Frame: at base line, 1 month and 3 months after treatment]
probing depth | [Time Frame: at base line, 1 month and 3 months after treatment]
  The measurement will be recorded by UNC15(University of North Carolina) periodontal probe . Pocket depth will be measured as the distances from the free gingival margin to the base of the periodontal pocket.

SECONDARY OUTCOMES:
-Plaque index (PI) | [Time Frame: at base line, 1 month and 3 months after treatment]
  It used to assess plaque accumulation around gingival margin.
  The degree of plaque accumulation was recorded as follow:
  * 0= No plaque around the gingival margin.
  * 1= A thin film of plaque around the gingival margin. The plaque may be recognized only by running a probe across the tooth surface.
  * 2= Moderate accumulation of soft deposits on the gingival margin and/or adjacent tooth surface, which can be seen by naked eye. 3= Abundance plaque accumulation within the gingival pocket and/or on the gingival margin and adjacent tooth surface and hard deposits on the tooth surface are seen.
Gingival index (GI) | [Time Frame: at base line, 1 month and 3 months after treatment]
  It used to assess gingival inflammation. The degree of gingival inflammation will be recorded as follow:
  * 0 = Normal gingiva.
  * 1 = Mild inflammation, slight change in color, slight edema and no bleeding on probing.
  * 2= Moderate inflammation, redness, edema and bleeding on probing.
  * 3= Severe inflammation, marked redness, edema and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mortada Fikry, professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: reatment of 3-wall intrabony defects in patients with chronic periodontitis with autologous platelet-rich fibrin: A randomized controlled clinical trial. J — https://scholar.google.com/scholar?output=instlink&q=info:gs7OSorwlysJ:scholar.google.com/&hl=ar&as_sdt=0,5&scillfp=3380595959201488678&oi=lle
- See also: Clinical significance of non-surgical periodontal therapy: an evidence-based perspective of scaling and root planing — https://scholar.google.com/scholar?output=instlink&q=info:XGpLL_1qxLQJ:scholar.google.com/&hl=ar&as_sdt=0,5&scillfp=2796192741746260869&oi=lle
- See also: Regeneration of periodontal intrabony defects using platelet-rich fibrin (PRF): A systematic review and network meta-analysis. Odontology — https://link.springer.com/content/pdf/10.1007/s10266-024-00949-7.pdf
- See also: Strategies of cell and cell-free therapies for periodontal regeneration: the state of the art. — https://link.springer.com/content/pdf/10.1186/s13287-022-03225-z.pdf